CLINICAL TRIAL: NCT00845338
Title: A 4-week, Open-label, Multicenter, Urodynamic Pilot Study to Explore the Efficacy, Tolerability and Safety of Darifenacin (7.5 mg With Up-titration to 15 mg) in Patients With Multiple Sclerosis and Neurogenic Detrusor Overactivity
Brief Title: Study of Darifenacin in Patients Suffering From Multiple Sclerosis and Neurogenic Detrusor Overactivity
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The enrollment rate at most centers was unlikely to result in the recruitment of the planned sample size of 40 evaluable subjects.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12331; 2006-002361-39 (EudraCT Number)
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Multiple Sclerosis; Overactive Detrusor
Keywords: Darifenacin; Multiple Sclerosis; Open Label Study
MeSH Terms: conditions — Multiple Sclerosis; Urinary Bladder, Overactive | interventions — darifenacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Darifenacin (BAY79-4998)

INTERVENTIONS:
Drug: Darifenacin (BAY79-4998) — Darifenacin 7,5mg tablets once daily for 14 days, darifenacin 7,5mg or 15mg once daily for 14 consecutive days

SUMMARY:
The objective of this study is to explore the effects of darifenacin in patients with multiple sclerosis and neurogenic detrusor overactivity. The efficacy, safety and tolerability of darifenacin are already well established in idiopathic detrusor overactivity. Patients with multiple sclerosis and neurogenic detrusor overactivity without detrusor-sphincter-dyssynergia (DSD) will be allocated to darifenacin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple sclerosis for at least 6 months
* Neurogenic detrusor overactivity without DSD
* Symptoms of OAB
* Patients capable of completing the bladder diary
* Patients capable of independent toileting
* Patients able to swallow the study medication in accordance to the protocol
* Body Mass Index >/= 18,8 kg/qm and </= 35,0 kg/qm
* documented, dated, written informed consent

Exclusion Criteria:

* Treatment with drugs known to affect mainly the urinary function 14 days prior to starting completion of the baseline diary for Visit 2
* Participation in a bladder-training program
* Low compliance bladder (Compliance <20 mL/cm H2O)
* DSD, Detrusor hyporeflexia / areflexia and bradykinesia / tremor of the external urethral sphincter
* Indwelling catheter or intermittent self-catheterization
* Patience with post-void residual (PVR) urinary volume > 200 mL at baseline
* Urinary retention or clinically significant bladder outlet obstruction as detected by the investigator
* Clinically predominant and bothersome stress urinary incontinence
* Neurological diseases other than multiple sclerosis affecting urinary bladder function
* Any urogenital surgery within 12 month prior to Visit 1
* 17 Additional Exclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in volume at first detrusor contraction as determined by urodynamics | At week 4

SECONDARY OUTCOMES:
Detrusor pressure at first contraction | At week 4
Volume at first detectable leakage | At week 4
Volume at 10/20/30/40 cm H2O | At week 4
Compliance | At week 4
Maximum cystometric bladder capacity | At week 4
7-day micturition diary: Micturitions | At days 0, 14, 28
7-day micturition diary: Urgency episodes | At days 0, 14, 28
7-day micturition diary: Urge urinary incontinence episodes | At days 0, 14, 28

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (15):
- Germany (15):
  - Emmendingen, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Lahr, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Villingen-Schwenningen, Baden-Wurttemberg
  - Planegg, Bavaria
  - Hamburg, Hamburg
  - Oberursel, Hesse
  - Herne, North Rhine-Westphalia
  - Mönchengladbach, North Rhine-Westphalia
  - Mülheim, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Halle, Saxony-Anhalt
  - Berlin, State of Berlin
  - Bad Berka, Thuringia

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/